CLINICAL TRIAL: NCT01661894
Title: Effectiveness of a Brain-Computer Interface Based System for Cognitive Enhancement in the Normal Elderly
Acronym: 3ECog
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Agency for Science, Technology and Research (Other); National University of Singapore (Other); Singapore Clinical Research Institute (Other); Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Lee Tih Shih, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-363
Record Dates: First submitted 2012-05-17; First posted 2012-08-10 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Age-Related Cognitive Decline; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Subjects will undergo the BrainpalTM intervention for 24 sessions over the span of 8 weeks. Each session will take 30-minute to complete. The intervention group will undergo the BrainpalTM treatment in the first 8 weeks of the trial.
  Interventions: Device: BrainPalTM
- Wait-List Control (No Intervention): The waitlist control will start their 8 week treatment after the completion of the intervention group from week 9 onwards. They will undergo the BCI intervention for 24 sessions over the span of 8 weeks.

INTERVENTIONS:
Device: BrainPalTM — Brain-computer Interface (BCI) is a direct communication pathway between a human brain and an external device. It is a technology that enables people to interact with computers through their thoughts. Electroencephalography (EEG) is the best studied non-invasive interface facilitating such communication. The BCI system will take EEG recordings from the prefrontal cortex to determine the participants' state of attention with high specificity. The training program developed using this patented technology may be useful for individuals who experience difficulty with memory and sustaining their attention.
  Other Names: Brain-Computer Interface
  Arms: Intervention

SUMMARY:
The primary objective is to examine the efficacy of 8-weeks of a locally developed brain-computer interface based system (BrainpalTM)intervention for improving attention and memory in normal elderly. We hypothesize that elderly who have completed the training program will have significant improvement in their attention and memory compared to the controls, based on the Repeatable Battery for the Assessment of Neuropsychological Status.

DETAILED DESCRIPTION:
The world population has reached an unprecedented seven billion, with global population ageing increasing at a greater rate than total population growth. Between 1998 and 2030, the proportion of persons aged 65 years and over in Singapore will grow by about 3% annually compared to 1.0-1.3% in some developed nations. Specific cognitive deficits like inattention, dysexecutive functioning, and processing speed decline may affect a number of quality of life domains. Concurrent with these statistics, the maintenance of the highest possible level of cognitive functioning for as long as possible has become an important goal of aging successfully.

To contribute to the realization of this goal we propose to conduct a wait-list control pilot trial to examine the efficacy and safety of BrainpalTM for cognitive enhancement in the normal elderly. BrainpalTM uses a technology which analyzes brain waves captured through an electroencephalogram to determine the participants' state of attention. The training program developed using this patented technology may be useful for individuals who experience difficulty with memory and sustaining their attention.

BrainpalTM may represent one alternative means to enhance cognitive abilities and to slow down cognitive decline in the normal elderly. If demonstrated to be efficacious, this therapy may even help to delay the onset of dementia.

In addition, the rate of cognitive decline during the course of AD is possibly influenced by not only environmental but also genetic factors. To date, several genes, such as apolipoprotein E (APOE) and TOMM40 (translocase of outer mitochondrial membrane 40 homologue), have been identified to be probable genetic risk markers for AD. These genes have been shown to play a role in disease onset as well as rates of cognitive decline. For instance, studies have shown APOEε4 allele carriers to be associated with earlier and faster cognitive decline.

Therefore, we propose to analyse if there is any relationship between the genetic profiles of our participants and their performance in the BrainpalTM training program.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 60-70 years old
2. Clinical Dementia Rating (CDR) of 0.5*
3. Geriatric Depression Scale (GDS) of 9 and below
4. Mini-Mental State Examination of 24 and above*
5. Chinese ethnicity
6. Literate in English and/or Chinese
7. Able to travel to study site independently

   * In the case of conflicting CDR and MMSE scores, MMSE scores will supersede CDR scores.

Exclusion Criteria:

1. Any known neuropsychiatric disorders (such as epilepsy or mental retardation)
2. Involvement in another research study (aside from SLAS)

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Total Score on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Comparison in the change of RBANS total score from baseline (Week 1) to post-treatment (Week 8) in Intervention Group versus Wait-List Control group
  The Total Score on RBANS reflects the neurocognitive status of the participant by summing five index/domain scores. The domains are Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory.

SECONDARY OUTCOMES:
Number of Adverse Events reported by participants on the Safety Measurement Form | The duration of 8 weeks of intensive BCI intervention sessions
  The Safety Measurement Form will be completed at the start of every BCI intervention visit (except the first visit). It will collect information on any safety concerns and/or side effects experienced by the participant since their last BCI intervention visit.
Usability Measurement | Before a subject exits from the study, including completion of the protocol and withdraw of consent
  The usability measurement collects feedback on the acceptability and usability of the BCI intervention program to improve user satisfaction in future trials.

OTHER OUTCOMES:
Relationship between genetic profile of participants and their performance on the BrainpalTM training program | After the BrainpalTM training program is completed
  Blood samples will be collected from each subject for DNA extraction. The samples will be used to generate a genetic profile for each subject. The presence or absence of genes of interest (i.e. TOMM40 and APOEε4)on a subject's genetic profile will then be associated with his or her corresponding performance on BCI, as measured by his or her RBANS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Tih Shih Lee, MD, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Lee TS, Goh SJ, Quek SY, Phillips R, Guan C, Cheung YB, Feng L, Teng SS, Wang CC, Chin ZY, Zhang H, Ng TP, Lee J, Keefe R, Krishnan KR. A brain-computer interface based cognitive training system for healthy elderly: a randomized control pilot study for usability and preliminary efficacy. PLoS One. 2013 Nov 18;8(11):e79419. doi: 10.1371/journal.pone.0079419. eCollection 2013. PMID 24260218